CLINICAL TRIAL: NCT01247753
Title: Stepping Up to Health - Walking Exercise and Nutrition to Reduce Diabetes Risk for You (WENDY)
Brief Title: Walking Exercise and Nutrition to Reduce Diabetes Risk for You (WENDY)
Acronym: WENDY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Mater Mothers' Hospital (Other)
Responsible Party: Principal Investigator, Catherine Kim, associate professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K23 DK71552-1; K23DK071552 (NIH)
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Diabetes; Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Walking group
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Walking group — Internet-mediated pedometer-based walking program with gradually increasing step count goals and feedback on step counts. Also includes nutritional coaching course consisting of 1 individual session with a dietician, 4 group sessions, and monthly follow-up. Oral glucose tolerance tests pre and post-intervention.
  Arms: Intervention

SUMMARY:
The prevalence of Gestational Diabetes Mellitus (GDM) in Australia is approximately 5%-8%, with up to one third of all parous women who develop type 2 diabetes having a previous history of GDM. Research to determine strategies to delay or prevent the development of or progression to diabetes is vital, particularly in population groups that are at higher risk, such as GDM, and overweight women (BMI>=25). Currently, follow-up or post-partum support for women who develop GDM is limited to advice to complete a 6 week post-partum oral glucose tolerance test to exclude overt diabetes, to be repeated annually. A pilot randomized controlled trial (RCT) conducted at Mater Mothers Hospital suggested that a post-partum intervention designed to increase physical activity in women with previous GDM may be feasible. A recent study in the United States recruited women with recent GDM into an RCT where the control group received usual care and the intervention group received a web based walking program. Although the results of this study are limited, they did show an increase in pedometer steps/day between baseline and end of study. Dietary intervention has been proven to increase probability of weight loss, so a strategy of combining both a pedometer and nutrition based program may prove to be more successful for long term improvement of a healthy lifestyle to prevent type 2 diabetes.

Study hypothesis: A pedometer based intervention to encourage physical activity, combined with nutrition coaching in women with recent GDM and BMI >= 25 will result in increased weight loss, improved insulin sensitivity and increased physical activity when compared with standard care.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of gestational diabetes mellitus and given birth in the preceding 6 months to 3 years; 18 years of age or older; BMI >= 25; Routine access to a computer; Adequate computer skills to navigate websites and email; Speak and understand English well enough to participate in the study

Exclusion Criteria:

Currently pregnant or planning to become pregnant in the next year; Current diabetes; Currently taking medications that interfere with glucose metabolism

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2012-03-01 (Actual); Study Completion 2012-03-01 (Actual)

PRIMARY OUTCOMES:
Change in body weight | pre-post

SECONDARY OUTCOMES:
Change in insulin sensitivity | pre-post
Change in physical activity | pre-post

CONTACTS AND LOCATIONS:
Locations (1):
- Mater Mothers Hospital, South Brisbane, Queensland, Australia